CLINICAL TRIAL: NCT06512272
Title: Evaluating Feasibility and Acceptability of Video Discharge Hosted in Patient Knows Best or Ortus-iHealth Apps: A Feasibility Randomised Controlled Trial
Brief Title: Video-recOrded hospItal dischaRge (VOIR)
Acronym: VOIR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Collaborators: Basildon and Thurrock Hospitals NHS FoundationTrust (Unknown); Southend NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 320936; 423607 (Other: 423607)
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-03

CONDITIONS: ALL, Adult
Keywords: hospital discharge; video recorded discharge; transition of care; mobile application
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Randomisation on a ratio of 1:1
  * A: allocated usual care
  * B: allocated intervention group which include usual care plus video-recorded discharge
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Usual hospital discharge include medical discharge letter and verbal advice from healthcare team.
- Intervention group (Other): Usual hospital discharge + video recorded medical advice from the healthcare team uploaded in a mobile app
  Interventions: Other: Video recorded shared using a mobile application

INTERVENTIONS:
Other: Video recorded shared using a mobile application — The routine hospital discharge explanation is video recorded [up to three minutes].
  The video is uploaded by to a mobile app for the patient and patient/ relatives can review the advice multiple times
  Arms: Intervention group

SUMMARY:
This study evaluates the suitability and acceptability of video-recorded discharge via the Patient Knows Best app. Through a randomized control trial, patients receive either standard discharge care or standard care supplemented with video-recorded discharge. Clinical teams record briefings covering medication and wound care, which patients can access multiple times on their smart devices. Patients and clinical staff complete questionnaires to assess acceptance and feasibility. Feasibility is determined by recruitment, retention, and completion rates, with patient engagement and viewing habits also analyzed. The study aims to enhance patient understanding and continuity of care through accessible discharge information.

DETAILED DESCRIPTION:
Study Design

The study aims to assess how suitable and acceptable the use of video-recorded discharge via the Patient Knows Best or Ortus-iHealth application is. It employs a randomised control trial design, with one group receiving standard discharge care and another receiving the standard care plus video-recorded discharge.

Upon discharge from hospital, the clinical team (e.g, nurses and doctors) will record the routine discharge briefing, covering aspects such as medication and wound care, for consenting patients. This briefing will be based on the discharge letter from the medical team and will last approximately up to three minutes. It will take place in a private hospital ward room, using the patient's or their relative's smart device (e.g., mobile or tablet). Subsequently, the recorded video will be uploaded to the patient's Patient Knows Best app account. Patients can review the video multiple times to reinforce their understanding of the discharge information, including medication advice, wound dressing, and exercise. Additionally, they can share it with their relatives, as well as community and district nursing teams, to enhance the clarity of shared information and continuity of care.

Both control and intervention group patients will receive a self-reported questionnaire regarding their acceptance of the discharge process, satisfaction levels, and its impact on their quality of life. Clinical staff involved in the recording will also complete a questionnaire assessing the feasibility, practicality, and satisfaction with the new intervention.

The feasibility of the study will be evaluated based on recruitment numbers, retention rates, completion rates, and the chosen questionnaire's suitability. Questionnaires will be administered post-discharge, one week after discharge, and thirty days later. Additionally, patient engagement with the Patient Knows Best platform and video viewing habits will be analysed to explore any differences among demographic groups.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Anticipated to be discharged to their own home or that of a relative;
* Staying for at least one night on a participating hospital ward;
* Recently discharge (in the last 2 months) from the participating hospital ward with the same clinical problem as assessed by the care professionals;
* From cardiothoracic centre-Basildon or Elderly ward-Southend
* Have a personal digital device (e.g., mobile or tablet)/ or their close relative and mobile app
* Able to read and understand English.
* Relative or patient willing and able to give informed consent
* Clinical Frailty scale of ≤ 8 using Rockwood Frailty Scale

Exclusion Criteria:

* Patients live out of the area or plan to be transferred to another acute hospital;
* Discharged after recurrent admissions for the same clinical complaint as assessed by the care professionals;
* Patient or immediate carer don't have a personal digital device capable of hosting Patient Knows Best/ Ortus-iHealth app;
* Patient or relative unable or unwilling to upload the personalised discharge video to mobile app;
* Admitted for psychiatric reasons (other than dementia/delirium);
* Identified as being at the end of life and whose care has become palliative / clinical Frailty scale of > 8 using Rockwood Frailty Scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of video-discharge | 7 days and 30 days post-discharge
  Questionnaire with close ended and open ended question based on validated questionnaire

SECONDARY OUTCOMES:
Patient satisfaction | 7 and 30 days post discharge
  Brief questionnaire on patient satisfaction
Care of Transitions | 7 and 30 days post discharge
  Three questions measuring validated tool
Staff satisfaction of video recorded discharge | within 7 days of post-discharge experience
  Close and opened questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Naim Abdulmohdi, PhD, Principal Investigator — Anglia Ruskin University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barker RE, Jones SE, Banya W, Fleming S, Kon SSC, Clarke SF, Nolan CM, Patel S, Walsh JA, Maddocks M, Farquhar M, Bell D, Wedzicha JA, Man WD. The Effects of a Video Intervention on Posthospitalization Pulmonary Rehabilitation Uptake. A Randomized Controlled Trial. Am J Respir Crit Care Med. 2020 Jun 15;201(12):1517-1524. doi: 10.1164/rccm.201909-1878OC. PMID 32182098
- [Background] Baxter R, Murray J, Cockayne S, Baird K, Mandefield L, Mills T, Lawton R, Hewitt C, Richardson G, Sheard L, O'Hara JK; PACT research team. Improving the safety and experience of transitions from hospital to home: a cluster randomised controlled feasibility trial of the 'Your Care Needs You' intervention versus usual care. Pilot Feasibility Stud. 2022 Oct 1;8(1):222. doi: 10.1186/s40814-022-01180-3. PMID 36183129
- [Background] Forster AJ, Murff HJ, Peterson JF, Gandhi TK, Bates DW. The incidence and severity of adverse events affecting patients after discharge from the hospital. Ann Intern Med. 2003 Feb 4;138(3):161-7. doi: 10.7326/0003-4819-138-3-200302040-00007. PMID 12558354
- [Background] Hesselink G, Schoonhoven L, Barach P, Spijker A, Gademan P, Kalkman C, Liefers J, Vernooij-Dassen M, Wollersheim H. Improving patient handovers from hospital to primary care: a systematic review. Ann Intern Med. 2012 Sep 18;157(6):417-28. doi: 10.7326/0003-4819-157-6-201209180-00006. PMID 22986379
- [Background] Hoek AE, Joosten M, Dippel DWJ, van Beeck EF, van den Hengel L, Dijkstra B, Papathanasiou D, van Rijssel D, van den Hamer M, Schuit SCE, Burdorf A, Haagsma JA, Rood PPM. Effect of Video Discharge Instructions for Patients With Mild Traumatic Brain Injury in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2021 Mar;77(3):327-337. doi: 10.1016/j.annemergmed.2020.10.023. PMID 33618811
- [Background] Kapoor A, Field T, Handler S, Fisher K, Saphirak C, Crawford S, Fouayzi H, Johnson F, Spenard A, Zhang N, Gurwitz JH. Adverse Events in Long-term Care Residents Transitioning From Hospital Back to Nursing Home. JAMA Intern Med. 2019 Sep 1;179(9):1254-1261. doi: 10.1001/jamainternmed.2019.2005. PMID 31329223
- [Background] Le Berre M, Maimon G, Sourial N, Gueriton M, Vedel I. Impact of Transitional Care Services for Chronically Ill Older Patients: A Systematic Evidence Review. J Am Geriatr Soc. 2017 Jul;65(7):1597-1608. doi: 10.1111/jgs.14828. Epub 2017 Apr 12. PMID 28403508
- [Background] Laugaland K, Aase K, Barach P. Interventions to improve patient safety in transitional care--a review of the evidence. Work. 2012;41 Suppl 1:2915-24. doi: 10.3233/WOR-2012-0544-2915. PMID 22317162
- [Background] Mallet KH, Shamloul RM, Lecompte-Collin J, Winkel J, Donnelly B, Dowlatshahi D. Telerehab at Home: Mobile Tablet Technology for Patients With Poststroke Communication Deficits-A Pilot Feasibility Randomized Control Trial. J Speech Lang Hear Res. 2023 Feb 13;66(2):648-655. doi: 10.1044/2022_JSLHR-21-00616. Epub 2023 Jan 12. PMID 36634230
- [Background] Wang Q, Lee RL, Hunter S, Chan SW. Patients' experiences of using a mobile application-based rehabilitation programme after total hip or knee arthroplasty: a qualitative descriptive study. BMC Nurs. 2023 Jul 27;22(1):246. doi: 10.1186/s12912-023-01409-3. PMID 37496003